CLINICAL TRIAL: NCT05201859
Title: A Randomized, Open-Label, Phase II Study to Evaluate the Efficacy and Safety of Sintilimab Plus Capecitabine Versus Capecitabine Alone as Adjuvant Therapy for Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Adjuvant Sintilimab Plus Capecitabine in Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-486
Record Dates: First submitted 2022-01-20; First posted 2022-01-21 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab; spartalizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Sintilimab Plus Capecitabine (Experimental): Lead-in Phase: Sintilimab (200mg, D1, D14 for 2 cycles); Adjuvant Phase: Sintilimab ( 200mg D1, every three weeks, a total of 24 weeks, 8 cycles) + Capecitabine ( 1000 mg/m2, BID, D1-14 every three weeks, a total of 24 weeks, 8 cycles).
  Interventions: Drug: Sintilimab; Drug: Capecitabine
- Adjuvant Capecitabine (Active Comparator): Capecitabine 1000 mg/m2, BID, D1-14, every three weeks, a total of 24 weeks, 8 cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Sintilimab — Sintilimab is a humanized monoclonal antibody against Programmed death 1(PD-1).
  Other Names: Anti-PD-1 Antibody; IBI308
  Arms: Adjuvant Sintilimab Plus Capecitabine
Drug: Capecitabine — An oral anticancer agent that can be converted into 5-Fu in vivo.

SUMMARY:
This randomized clinical trial determining whether Sintilimab plus Capecitabine versus Capecitabine alone can improve the progression-free survival rate of NPC patients with unfavorable response to induction chemotherapy. Patients whose plasma EBV DNA> 0 copy/mL or SD/PD according to RECIST1.1 after two cycles induction chemotherapy will have concurrent chemoradiotherapy. MRI, CT and EBV DNA will be assessed before the end of radiotherapy. After concurrent chemoradiotherapy, eligible patients will be randomized to receive either adjuvant Sintilimab plus Capecitabine or Capecitabine alone.

DETAILED DESCRIPTION:
Currently, although NCCN (National Comprehensive Cancer Network) guidelines recommend induction chemotherapy combined with concurrent chemoradiotherapy as IIA level-evidenced treatment for nasopharyngeal carcinoma (NPC), there are still about 20-30% of patients with NPC who experienced recurrence and metastasis after radical treatment.

Our previous results showed that patients with plasma Epstein-Barr virus (EBV) DNA > 0 copy/mL or stable disease/progressive disease (SD/PD) after induction chemotherapy had a significantly higher risk of disease progression than patients with plasma EBV DNA=0 copy/mL and complete response/partial response (CR/PR), according to Response Evaluation Criteria in Solid Tumors (RECIST). As for these high-risk patients, the urgent clinical problem to be solved is whether increased adjuvant treatment intensity after concurrent chemoradiotherapy can improve their survival rates.

The addition of adjuvant capecitabine to chemoradiotherapy significantly improved survival in patients with NPC, with a manageable safety profile. Sintilimab is a humanized monoclonal antibody against programmed death 1(PD-1). Anti-PD-1 monoclonal antibody showed efficacy and safety in previous studies, however, the efficacy of immunotherapy alone was limited. Several prospective studies have shown that anti-PD-1 monoclonal antibody combined with chemotherapy had a synergistic effect.

Based on this, this randomized clinical trial determining whether adjuvant Sintilimab plus Capecitabine versus Capecitabine alone can improve the progression-free survival rate of patients with unfavorable response to induction chemotherapy and may provide new evidence for individualized comprehensive treatment of NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III.
2. Tumor staged as II-IVa (AJCC 8th,excluding T2N0 disease).
3. Age ≥ 18 years and ≤ 70 years, both genders.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
5. Patients with plasma EBV DNA> 0 copy/mL or PD/SD according to RECIST1.1 after two cycles of induction chemotherapy.
6. Completed protocol-specified curative chemoradiotherapy, including two cycles of induction chemotherapy, intensity-modulated radiotherapy, and concurrent cisplatin chemotherapy( at least 2 cycles of concurrent cisplatin chemotherapy).
7. Completion of the last radiation dose within 1 to 7 days before randomization
8. No progression after prior cCRT
9. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
10. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
11. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
12. Patients must be informed of the investigational nature of this study and give written informed consent.
13. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I).
2. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
3. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
4. Is pregnant or breastfeeding.
5. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml
6. Hepatitis C virus (HCV) antibody positive
7. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
8. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
9. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
10. Has known allergy to large molecule protein products or any compound of sintilimab.
11. Has a known history of interstitial lung disease.
12. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  Defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Defined as the time from random assignment to death from any cause or censored at the date of last follow-up
Locoregional Relapse-Free Survival (LRFS) | 2 years
  Defined as the time from random assignment to local or regional relapse, or death from any cause.
Distant Metastasis-Free Survival (DMFS) | 2 years
  Defined as the time from random assignment to distant metastasis, or death from any cause.
Incidence rate of adverse events (AEs) | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Lee AW, Lau WH, Tung SY, Chua DT, Chappell R, Xu L, Siu L, Sze WM, Leung TW, Sham JS, Ngan RK, Law SC, Yau TK, Au JS, O'Sullivan B, Pang ES, O SK, Au GK, Lau JT; Hong Kong Nasopharyngeal Cancer Study Group. Preliminary results of a randomized study on therapeutic gain by concurrent chemotherapy for regionally-advanced nasopharyngeal carcinoma: NPC-9901 Trial by the Hong Kong Nasopharyngeal Cancer Study Group. J Clin Oncol. 2005 Oct 1;23(28):6966-75. doi: 10.1200/JCO.2004.00.7542. PMID 16192584
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Liu LT, Tang LQ, Chen QY, Zhang L, Guo SS, Guo L, Mo HY, Zhao C, Guo X, Cao KJ, Qian CN, Zeng MS, Bei JX, Hong MH, Shao JY, Sun Y, Ma J, Mai HQ. The Prognostic Value of Plasma Epstein-Barr Viral DNA and Tumor Response to Neoadjuvant Chemotherapy in Advanced-Stage Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2015 Nov 15;93(4):862-9. doi: 10.1016/j.ijrobp.2015.08.003. Epub 2015 Aug 7. PMID 26530755
- [Background] Bonner JA, Harari PM, Giralt J, Cohen RB, Jones CU, Sur RK, Raben D, Baselga J, Spencer SA, Zhu J, Youssoufian H, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for locoregionally advanced head and neck cancer: 5-year survival data from a phase 3 randomised trial, and relation between cetuximab-induced rash and survival. Lancet Oncol. 2010 Jan;11(1):21-8. doi: 10.1016/S1470-2045(09)70311-0. Epub 2009 Nov 10. PMID 19897418
- [Background] Tao Y, Auperin A, Sun X, Sire C, Martin L, Coutte A, Lafond C, Miroir J, Liem X, Rolland F, Even C, Nguyen F, Saada E, Maillard A, Colin-Batailhou N, Thariat J, Guigay J, Bourhis J. Avelumab-cetuximab-radiotherapy versus standards of care in locally advanced squamous-cell carcinoma of the head and neck: The safety phase of a randomised phase III trial GORTEC 2017-01 (REACH). Eur J Cancer. 2020 Dec;141:21-29. doi: 10.1016/j.ejca.2020.09.008. Epub 2020 Oct 24. PMID 33125944
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Chen YP, Liu X, Zhou Q, Yang KY, Jin F, Zhu XD, Shi M, Hu GQ, Hu WH, Sun Y, Wu HF, Wu H, Lin Q, Wang H, Tian Y, Zhang N, Wang XC, Shen LF, Liu ZZ, Huang J, Luo XL, Li L, Zang J, Mei Q, Zheng BM, Yue D, Xu J, Wu SG, Shi YX, Mao YP, Chen L, Li WF, Zhou GQ, Sun R, Guo R, Zhang Y, Xu C, Lv JW, Guo Y, Feng HX, Tang LL, Xie FY, Sun Y, Ma J. Metronomic capecitabine as adjuvant therapy in locoregionally advanced nasopharyngeal carcinoma: a multicentre, open-label, parallel-group, randomised, controlled, phase 3 trial. Lancet. 2021 Jul 24;398(10297):303-313. doi: 10.1016/S0140-6736(21)01123-5. Epub 2021 Jun 7. PMID 34111416
- [Background] Meric-Bernstam F, Larkin J, Tabernero J, Bonini C. Enhancing anti-tumour efficacy with immunotherapy combinations. Lancet. 2021 Mar 13;397(10278):1010-1022. doi: 10.1016/S0140-6736(20)32598-8. Epub 2020 Dec 4. PMID 33285141
- [Background] Yang S, Haluska FG. Treatment of melanoma with 5-fluorouracil or dacarbazine in vitro sensitizes cells to antigen-specific CTL lysis through perforin/granzyme- and Fas-mediated pathways. J Immunol. 2004 Apr 1;172(7):4599-608. doi: 10.4049/jimmunol.172.7.4599. PMID 15034078
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578